CLINICAL TRIAL: NCT02011490
Title: An Open-Label, Single-Dose Study to Investigate the Pharmacokinetics of MK-8616 in Subjects With Moderate and Severe Renal Insufficiency
Brief Title: Pharmacokinetics of Sugammadex (MK-8616) in Participants With Moderate and Severe Renal Insufficiency (MK-8616-105)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8616-105
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Results first posted 2015-02-10 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Renal Insufficiency; Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — Sugammadex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Severe Renal Insufficiency Participants: Part 1 (Experimental): Participants with severe renal insufficiency will receive a single dose of 4 mg/kg sugammadex administered as an IV bolus over 10 seconds. Dose will be administered by direct injection into a peripheral vein.
  Interventions: Drug: sugammadex
- Moderate Renal Insufficiency Participants: Part 1 (Experimental): Participants with moderate renal insufficiency will receive a single dose of 4 mg/kg sugammadex administered as an IV bolus over 10 seconds. Dose will be administered by direct injection into a peripheral vein.
  Interventions: Drug: sugammadex
- Healthy Control Participants: Part 1 (Experimental): Healthy control participants will receive a single dose of 4 mg/kg sugammadex administered as an IV bolus over 10 seconds. Dose will be administered by direct injection into a peripheral vein.
  Interventions: Drug: sugammadex
- Severe Renal Insufficiency Participants: Part 2 (Experimental): Participants with severe renal insufficiency will receive a single dose of 4 mg/kg sugammadex administered as an IV bolus over 10 seconds. Dose will be administered into a peripheral vein through an IV catheter connected to an IV tubing with injection port. The IV tubing is connected to a saline bag. Free-flowing access to the vein will be confirmed immediately prior to dose administration, and dose will be followed by saline flush.
  Interventions: Drug: sugammadex
- Moderate Renal Insufficiency Participants: Part 2 (Experimental): Participants with moderate renal insufficiency will receive a single dose of 4 mg/kg sugammadex administered as an IV bolus over 10 seconds. Dose will be administered into a peripheral vein through an IV catheter connected to an IV tubing with injection port. The IV tubing is connected to a saline bag. Free-flowing access to the vein will be confirmed immediately prior to dose administration, and dose will be followed by saline flush.
  Interventions: Drug: sugammadex
- Healthy Control Participants: Part 2 (Experimental): Healthy control participants will receive a single dose of 4 mg/kg sugammadex administered as an IV bolus over 10 seconds. Dose will be administered into a peripheral vein through an IV catheter connected to an IV tubing with injection port. The IV tubing is connected to a saline bag. Free-flowing access to the vein will be confirmed immediately prior to dose administration, and dose will be followed by saline flush.
  Interventions: Drug: sugammadex

INTERVENTIONS:
Drug: sugammadex — sugammadex 4 mg/kg IV bolus

SUMMARY:
The purpose of this study is to evaluate the plasma pharmacokinetics of a single 4 mg/kg intravenous (IV) dose of sugammadex in participants with moderate and severe renal insufficiency compared to that in participants with normal renal function. The study consists of two parts. In Part 1, participants with renal insufficiency and healthy participants will be administered study drug by IV bolus injection into a peripheral vein. In Part 2, participants with renal insufficiency and healthy participants will be administered study drug as an IV bolus into a peripheral vein, through an IV catheter connected to IV tubing with injection port. Subjects who participate in Part 1 of study may be enrolled in Part 2, which would reduce the overall number of participants enrolled for the study.

DETAILED DESCRIPTION:
In each study period (i.e., Part 1 and Part 2), day of drug administration was defined to be Day 1.

ELIGIBILITY:
Inclusion Criteria:

All Participants:

* Body Mass Index ≥18 to ≤40 kg/m^2
* Females of childbearing potential must either be sexually inactive (abstinent) for 14 days prior to dosing and throughout the study or are using an acceptable birth control method
* Females of non-childbearing potential must have undergone a sterilization procedure at least 6 months prior to dosing or are postmenopausal with amenorrhea for at least 1 year prior to dosing and have follicle stimulating hormone (FSH) serum levels consistent with postmenopausal status
* Male subjects must agree not to donate sperm from dosing until 90 days after dosing

Participants with Moderate or Severe Renal Insufficiency:

* Health of participant is stable based on medical history, laboratory tests and other assessments
* Clinical diagnosis of impaired stable renal function, and a creatinine clearance (CLcr) of <30 mL/min and not on hemodialysis for severe renal insufficiency participants, or 30 to <50 mL/min for moderate renal insufficiency participants
* No clinically significant change in renal status for at least 1 month prior to dosing, and is not currently or has not previously been on hemodialysis

Healthy Control Participants:

* Participant is medically healthy based on laboratory tests and other assessments
* Age of the individual healthy participants in Part 1 of the study is aimed to be within the range of the mean age ± approximately 15 years of all participants with renal impairment in Part 1 of the study combined; this approach will also be applied with respect to age of participants in Part 2 of the study
* CLcr ≥80 mL/min

Exclusion Criteria:

All Participants:

* Mentally or legally incapacitated, significant emotional problems at screening or expected during the conduct of the study or history of a clinically significant psychiatric disorder over the last 5 years
* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, or neurological disease whose current condition is considered unstable
* History or presence of alcoholism and drug abuse within the past 6 months
* History or presence of hypersensitivity or idiosyncratic reaction to the study medication or related compounds
* Female participants who are pregnant or lactating
* Positive results for the urine or saliva drug screen, or for the urine or breath alcohol screen
* Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV)
* Regular user of any medication (including over the counter) that would significantly alter renal function (e.g., cimetidine)
* Donation of blood or significant blood loss within 56 days prior to dosing, or donation of plasma within 7 days prior to dosing
* Participation in another clinical trial within 28 days prior to dosing
* No participant may be enrolled more than once within Part 1. Subjects who participate in Part 1 of study may be enrolled in Part 2, but participants within Part 2 are not to be enrolled more than once in Part 2

Healthy Control Participants:

* Participant has had a renal transplant or has had nephrectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-12-11 (Actual); Primary Completion 2014-06-06 (Actual); Study Completion 2014-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Investigational Site 001, Hialeah, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Min KC, Lasseter KC, Marbury TC, Wrishko RE, Hanley WD, Wolford DG, Udo de Haes J, Reitmann C, Gutstein DE. Pharmacokinetics of sugammadex in subjects with moderate and severe renal impairment . Int J Clin Pharmacol Ther. 2017 Sep;55(9):746-752. doi: 10.5414/CP203025. PMID 28679468
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=8616-105&kw=8616-105&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 33 subjects participated in study. 9 participated in both Part 1 and Part 2; for these, separate Part 2 baseline assessments were obtained. Due to differing Part 1 and Part 2 baseline renal function result, 1 participant was in severe renal insufficiency group in Part 1 and moderate renal insufficiency group in Part 2.
Groups:
- Severe Renal Insufficiency Participants: Part 1: Participants with severe renal insufficiency receive a single dose of 4 mg/kg sugammadex administered as an intravenous (IV) bolus over 10 seconds. In Part 1, dose is administered by direct injection into a peripheral vein.
- Moderate Renal Insufficiency Participants: Part 1: Participants with moderate renal insufficiency receive a single dose of 4 mg/kg sugammadex administered as an IV bolus over 10 seconds. In Part 1, dose is administered by direct injection into a peripheral vein.
- Healthy Control Participants: Part 1: Healthy control participants receive a single dose of 4 mg/kg sugammadex administered as an IV bolus over 10 seconds. In Part 1, dose is administered by direct injection into a peripheral vein.
- Severe Renal Insufficiency Participants: Part 2: Participants with severe renal insufficiency receive a single dose of 4 mg/kg sugammadex administered as an IV bolus over 10 seconds. In Part 2, dose is administered into a peripheral vein through an IV catheter connected to an IV tubing with injection port. The IV tubing is connected to a saline bag. Free-flowing access to the vein is confirmed immediately prior to dose administration, and dose is followed by saline flush.
- Moderate Renal Insufficiency Participants: Part 2: Participants with moderate renal insufficiency receive a single dose of 4 mg/kg sugammadex administered as an IV bolus over 10 seconds. In Part 2, dose is administered into a peripheral vein through an IV catheter connected to an IV tubing with injection port. The IV tubing is connected to a saline bag. Free-flowing access to the vein is confirmed immediately prior to dose administration, and dose is followed by saline flush.
- Healthy Control Participants: Part 2: Healthy control participants receive a single dose of 4 mg/kg sugammadex administered as an IV bolus over 10 seconds. In Part 2, dose administered into a peripheral vein through an IV catheter connected to an IV tubing with injection port. The IV tubing is connected to a saline bag. Free-flowing access to the vein is confirmed immediately prior to dose administration, and dose is followed by saline flush.
Period: Part 1
Arm/Group | Severe Renal Insufficiency Participants: Part 1 | Moderate Renal Insufficiency Participants: Part 1 | Healthy Control Participants: Part 1 | Severe Renal Insufficiency Participants: Part 2 | Moderate Renal Insufficiency Participants: Part 2 | Healthy Control Participants: Part 2
Started | 8 | 8 | 8 | 0 | 0 | 0
Completed | 8 | 8 | 8 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | Severe Renal Insufficiency Participants: Part 1 | Moderate Renal Insufficiency Participants: Part 1 | Healthy Control Participants: Part 1 | Severe Renal Insufficiency Participants: Part 2 | Moderate Renal Insufficiency Participants: Part 2 | Healthy Control Participants: Part 2
Started | 0 | 0 | 0 | 6 (4 had also participated in Part 1 (all in severe group)) | 6 (3 had also participated in Part 1 (2 in moderate, 1 in severe groups)) | 6 (2 had also participated in Part 1 (both in healthy group))
Completed | 0 | 0 | 0 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This table includes all 33 subjects who participated in study. Subjects who participated in both Part 1 and Part 2 are represented only once in this table. 1 participant was in severe renal insufficiency group in Part 1 and moderate renal insufficiency group in Part 2 and is allocated to severe renal insufficiency group in this table.
Groups:
- Severe Renal Insufficiency Participants: Part 1 + Part 2: This group includes participants with severe renal insufficiency who were included in Part 1, Part 2, or in both Part 1 and Part 2. Participants receive a single dose of 4 mg/kg sugammadex administered as an IV bolus over 10 seconds. In Part 1, dose is administered by direct injection into a peripheral vein. In Part 2, dose is administered into a peripheral vein through an IV catheter connected to an IV tubing with injection port.
- Moderate Renal Insufficiency Participants: Part 1 + Part 2: This group includes participants with moderate renal insufficiency who were included in Part 1, Part 2, or in both Part 1 and Part 2. Participants receive a single dose of 4 mg/kg sugammadex administered as an IV bolus over 10 seconds. In Part 1, dose is administered by direct injection into a peripheral vein. In Part 2, dose is administered into a peripheral vein through an IV catheter connected to an IV tubing with injection port.
- Healthy Control Participants: Part 1 + Part 2: This group includes healthy control participants who were included in Part 1, Part 2, or in both Part 1 and Part 2. Participants receive a single dose of 4 mg/kg sugammadex administered as an IV bolus over 10 seconds. In Part 1, dose is administered by direct injection into a peripheral vein. In Part 2, dose is administered into a peripheral vein through an IV catheter connected to an IV tubing with injection port.
- Total: Total of all reporting groups
Arm/Group | Severe Renal Insufficiency Participants: Part 1 + Part 2 | Moderate Renal Insufficiency Participants: Part 1 + Part 2 | Healthy Control Participants: Part 1 + Part 2 | Total
Number analyzed (Participants) | 10 | 11 | 12 | 33
Age, Continuous [Mean (Full Range); unit: Years] | 62.3 [47 to 76] | 64.2 [47 to 76] | 58.3 [50 to 67] | 61.5 [47 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 5 | 8
  Male | 8 | 10 | 7 | 25

OUTCOME MEASURES:

1. Primary Outcome: Geometric Least Squares Mean Area Under the Plasma Drug Concentration-time Curve From Time Zero to Infinity (AUC0-∞) Following a Single IV Dose of Sugammadex
Description: Plasma samples for determination of sugammadex pharmacokinetic parameters were obtained pre-dose and at specified post-dose time points. AUC0-∞ was calculated as the sum of the AUC to the last time point with a detectable plasma concentration (AUC0-last, determined by trapezoidal method) and the extrapolated area given by Cest,last/λz, where Cest,last is the estimated concentration corresponding to the time of the last measurable concentration and λz is the apparent first-order terminal elimination rate constant. For each subject, λz was calculated by regression of the terminal log-linear portion of the plasma concentration-time profile. The reported least squares mean is the geometric least squares mean, which is the back-transformed least squares mean from the analysis of variance (ANOVA) linear fixed-effect model performed on natural log-transformed values of AUC0-∞. This calculation also provides the associated 95% confidence interval.
Time Frame: For participants with: normal renal function - up to 48 hours post-dose (Part 1 + Part 2); moderate renal insufficiency - up to Day 28 (Part 1) or Day 10 (Part 2); severe renal insufficiency - up to Day 35 (Part 1) or Day 14 (Part 2)
Population: Pharmacokinetic analysis was performed only for Part 2 data for participants in Part 2. Analysis was not conducted for Part 1, as review of drug concentration data, and dosing issues noted at investigative sites, indicated that in some participants, doses may not have been administered directly into vein, and likely infiltrated surrounding tissue.
Measure: Least Squares Mean (95% Confidence Interval); unit: ug*hr/mL
Groups:
- Severe Renal Insufficiency Participants: Part 1: Participants with severe renal insufficiency receive a single dose of 4 mg/kg sugammadex administered as an IV bolus over 10 seconds. In Part 1, dose is administered by direct injection into a peripheral vein.
Arm/Group | Severe Renal Insufficiency Participants: Part 1 | Moderate Renal Insufficiency Participants: Part 1 | Healthy Control Participants: Part 1 | Severe Renal Insufficiency Participants: Part 2 | Moderate Renal Insufficiency Participants: Part 2 | Healthy Control Participants: Part 2
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 6
ug*hr/mL |  |  |  | 339 [268 to 428] | 151 [120 to 191] | 62.5 [49.5 to 79.0]
Statistical Analysis 1: Comparison: Severe Renal Insufficiency Participants: Part 2 vs Healthy Control Participants: Part 2; Log-transformed plasma values were modeled using an analysis of variance (ANOVA) linear fixed-effect model with population (severe insufficiency, moderate insufficiency, and healthy control) as a fixed effect; Test type: Superiority or Other; Geometric least squares mean ratio = 5.42, 90% CI 2-sided [4.12 to 7.11] — Difference in least squares means of log-transformed data (severe renal impaired - healthy) was back transformed to geometric least squares mean ratio (severe renal impaired/healthy)
Statistical Analysis 2: Comparison: Moderate Renal Insufficiency Participants: Part 2 vs Healthy Control Participants: Part 2; Log-transformed plasma values were modeled using an ANOVA linear fixed-effect model with population (severe insufficiency, moderate insufficiency, and healthy control) as a fixed effect; Test type: Superiority or Other; Geometric least squares mean ratio = 2.42, 90% CI 2-sided [1.84 to 3.17] — Difference in least squares means of log-transformed data (moderate renal impaired - healthy) was back transformed to geometric least squares mean ratio (moderate renal impaired/healthy)

2. Primary Outcome: Geometric Least Squares Mean Area Under the Plasma Concentration Versus Time Curve From Time Zero to the Last Measurable Concentration (AUC0-last) Following a Single IV Dose of Sugammadex
Description: Plasma samples for determination of sugammadex pharmacokinetic parameters were obtained pre-dose and at specified post-dose time points. AUC0-last was determined by trapezoidal method. The reported least squares mean is the geometric least squares mean, which is the back-transformed least squares mean from the ANOVA linear fixed-effect model performed on natural log-transformed values of AUC0-last. This calculation also provides the associated 95% confidence interval.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ug*hr/mL
Arm/Group | Severe Renal Insufficiency Participants: Part 1 | Moderate Renal Insufficiency Participants: Part 1 | Healthy Control Participants: Part 1 | Severe Renal Insufficiency Participants: Part 2 | Moderate Renal Insufficiency Participants: Part 2 | Healthy Control Participants: Part 2
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 6
ug*hr/mL |  |  |  | 335 [265 to 424] | 148 [117 to 187] | 61.1 [48.3 to 77.3]
Statistical Analysis 1: Comparison: Severe Renal Insufficiency Participants: Part 2 vs Healthy Control Participants: Part 2; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Geometric least squares mean ratio = 5.49, 90% CI 2-sided [4.18 to 7.22] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Moderate Renal Insufficiency Participants: Part 2 vs Healthy Control Participants: Part 2; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Geometric least squares mean ratio = 2.42, 90% CI 2-sided [1.84 to 3.18] — [estimate comment as in outcome 1, analysis 2]

3. Primary Outcome: Geometric Least Squares Mean Maximum Observed Plasma Concentration (Cmax) Following a Single IV Dose of Sugammadex
Description: Plasma samples for determination of sugammadex pharmacokinetic parameters were obtained pre-dose and at specified post-dose time points. Cmax was determined from the observed plasma concentration-time data. The reported least squares mean is the geometric least squares mean, which is the back-transformed least squares mean from the ANOVA linear fixed-effect model performed on natural log-transformed values of Cmax. This calculation also provides the associated 95% confidence interval.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | Severe Renal Insufficiency Participants: Part 1 | Moderate Renal Insufficiency Participants: Part 1 | Healthy Control Participants: Part 1 | Severe Renal Insufficiency Participants: Part 2 | Moderate Renal Insufficiency Participants: Part 2 | Healthy Control Participants: Part 2
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 6
ug/mL |  |  |  | 62.2 [50.2 to 77.1] | 60.6 [49.0 to 75.1] | 66.1 [53.3 to 81.8]
Statistical Analysis 1: Comparison: Severe Renal Insufficiency Participants: Part 2 vs Healthy Control Participants: Part 2; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Geometric least squares mean ratio = 0.94, 90% CI 2-sided [0.73 to 1.21] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Moderate Renal Insufficiency Participants: Part 2 vs Healthy Control Participants: Part 2; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Geometric least squares mean ratio = 0.92, 90% CI 2-sided [0.72 to 1.18] — [estimate comment as in outcome 1, analysis 2]

4. Primary Outcome: Geometric Mean Percent of AUC0-∞ That Was Extrapolated (AUC%Extrap) Following a Single IV Dose of Sugammadex
Description: Plasma samples for determination of sugammadex pharmacokinetic parameters were obtained pre-dose and at specified post-dose time points. AUC%extrap represents the percentage of the AUC0-∞ obtained by extrapolation, calculated as (1 - [AUC0-last/AUC0-∞]) multiplied by 100.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percent extrapolated
Arm/Group | Severe Renal Insufficiency Participants: Part 1 | Moderate Renal Insufficiency Participants: Part 1 | Healthy Control Participants: Part 1 | Severe Renal Insufficiency Participants: Part 2 | Moderate Renal Insufficiency Participants: Part 2 | Healthy Control Participants: Part 2
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 6
Percent extrapolated |  |  |  | 0.850 (43.5) | 2.14 (29.2) | 2.10 (45.3)

5. Primary Outcome: Geometric Mean Total Clearance (CL) Following a Single IV Dose of Sugammadex
Description: Plasma samples for determination of sugammadex pharmacokinetic parameters were obtained pre-dose and at specified post-dose time points. CL is a quantitative measure of the rate at which a drug substance is removed from the body, calculated as Dose/AUC0-∞.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Severe Renal Insufficiency Participants: Part 1 | Moderate Renal Insufficiency Participants: Part 1 | Healthy Control Participants: Part 1 | Severe Renal Insufficiency Participants: Part 2 | Moderate Renal Insufficiency Participants: Part 2 | Healthy Control Participants: Part 2
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 6
L/hr |  |  |  | 0.961 (26.8) | 2.27 (39.6) | 5.70 (16.0)

6. Primary Outcome: Geometric Mean Volume of Distribution During the Terminal Elimination Phase (Vz) Following a Single IV Dose of Sugammadex
Description: Plasma samples for determination of sugammadex pharmacokinetic parameters were obtained pre-dose and at specified post-dose time points. Vz was calculated as Dose/(AUC0-∞*λz).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Severe Renal Insufficiency Participants: Part 1 | Moderate Renal Insufficiency Participants: Part 1 | Healthy Control Participants: Part 1 | Severe Renal Insufficiency Participants: Part 2 | Moderate Renal Insufficiency Participants: Part 2 | Healthy Control Participants: Part 2
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 6
L |  |  |  | 18.3 (24.8) | 18.8 (24.2) | 20.4 (25.7)

7. Primary Outcome: Geometric Mean of Mean Residence Time (MRT) of Unchanged Drug in the Systemic Circulation Following a Single IV Dose of Sugammadex
Description: Plasma samples for determination of sugammadex pharmacokinetic parameters were obtained pre-dose and at specified post-dose time points. MRT is defined as the mean duration of time a drug molecule is present in the systemic circulation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Severe Renal Insufficiency Participants: Part 1 | Moderate Renal Insufficiency Participants: Part 1 | Healthy Control Participants: Part 1 | Severe Renal Insufficiency Participants: Part 2 | Moderate Renal Insufficiency Participants: Part 2 | Healthy Control Participants: Part 2
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 6
hr |  |  |  | 15.7 (26.2) | 7.02 (30.8) | 2.48 (13.4)

8. Primary Outcome: Geometric Mean Apparent Volume of Distribution Estimated at Steady-state (Vss) Following a Single IV Dose of Sugammadex
Description: Plasma samples for determination of sugammadex pharmacokinetic parameters were obtained pre-dose and at specified post-dose time points. Vss is the theoretical volume that the total amount of administered drug would have to occupy (if it were uniformly distributed), to provide the same concentration as it is in blood plasma at steady state, calculated as CL*MRT.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Severe Renal Insufficiency Participants: Part 1 | Moderate Renal Insufficiency Participants: Part 1 | Healthy Control Participants: Part 1 | Severe Renal Insufficiency Participants: Part 2 | Moderate Renal Insufficiency Participants: Part 2 | Healthy Control Participants: Part 2
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 6
L |  |  |  | 15.1 (19.7) | 15.9 (21.9) | 14.1 (20.4)

9. Primary Outcome: Median Time to Maximum Observed Plasma Concentration (Tmax) Following a Single IV Dose of Sugammadex
Description: Plasma samples for determination of sugammadex pharmacokinetic parameters were obtained pre-dose and at specified post-dose time points. Tmax was determined from the observed plasma concentration-time data.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hr
Arm/Group | Severe Renal Insufficiency Participants: Part 1 | Moderate Renal Insufficiency Participants: Part 1 | Healthy Control Participants: Part 1 | Severe Renal Insufficiency Participants: Part 2 | Moderate Renal Insufficiency Participants: Part 2 | Healthy Control Participants: Part 2
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 6
hr |  |  |  | 0.03 [0.03 to 0.08] | 0.03 [0.02 to 0.08] | 0.03 [0.03 to 0.08]

10. Primary Outcome: Median Time of the Last Measurable Plasma Concentration (Tlast) Following a Single IV Dose of Sugammadex
Description: Plasma samples for determination of sugammadex pharmacokinetic parameters were obtained pre-dose and at specified post-dose time points. Tlast was determined from the observed plasma concentration-time data.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hr
Arm/Group | Severe Renal Insufficiency Participants: Part 1 | Moderate Renal Insufficiency Participants: Part 1 | Healthy Control Participants: Part 1 | Severe Renal Insufficiency Participants: Part 2 | Moderate Renal Insufficiency Participants: Part 2 | Healthy Control Participants: Part 2
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 6
hr |  |  |  | 72.00 [71.99 to 143.99] | 24.00 [23.99 to 47.99] | 12.00 [11.99 to 12.00]

11. Primary Outcome: Geometric Mean Apparent First-order Terminal Elimination Half-life (t1/2) Following a Single IV Dose of Sugammadex
Description: Plasma samples for determination of sugammadex pharmacokinetic parameters were obtained pre-dose and at specified post-dose time points. Elimination t1/2 is the time it takes for the concentration of the drug in the body to decrease by half during the elimination phase, calculated as the natural log of 2 (ln[2])/λz.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Severe Renal Insufficiency Participants: Part 1 | Moderate Renal Insufficiency Participants: Part 1 | Healthy Control Participants: Part 1 | Severe Renal Insufficiency Participants: Part 2 | Moderate Renal Insufficiency Participants: Part 2 | Healthy Control Participants: Part 2
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 6
hr |  |  |  | 13.24 (35.50) | 5.73 (29.79) | 2.47 (13.49)

12. Primary Outcome: Geometric Mean Effective Half-life (t1/2eff) Following a Single IV Dose of Sugammadex
Description: Plasma samples for determination of sugammadex pharmacokinetic parameters were obtained pre-dose and at specified post-dose time points. t½eff was calculated as ln(2)*MRT.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Severe Renal Insufficiency Participants: Part 1 | Moderate Renal Insufficiency Participants: Part 1 | Healthy Control Participants: Part 1 | Severe Renal Insufficiency Participants: Part 2 | Moderate Renal Insufficiency Participants: Part 2 | Healthy Control Participants: Part 2
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 6
hr |  |  |  | 10.89 (26.15) | 4.87 (30.84) | 1.72 (13.36)

13. Primary Outcome: Geometric Mean Apparent First-order Terminal Elimination Rate Constant (λz) Following a Single IV Dose of Sugammadex
Description: Plasma samples for determination of sugammadex pharmacokinetic parameters were obtained pre-dose and at specified post-dose time points. λz was calculated by regression of the terminal log-linear portion of the plasma concentration-time profile.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hr
Arm/Group | Severe Renal Insufficiency Participants: Part 1 | Moderate Renal Insufficiency Participants: Part 1 | Healthy Control Participants: Part 1 | Severe Renal Insufficiency Participants: Part 2 | Moderate Renal Insufficiency Participants: Part 2 | Healthy Control Participants: Part 2
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 6
1/hr |  |  |  | 0.0524 (35.5) | 0.121 (29.8) | 0.280 (13.5)

ADVERSE EVENTS:
Time Frame: Up to Day 35 (Part 1) or Day 14 (Part 2)
Description: 33 subjects participated in study. 9 of these participated in both Part 1 and Part 2 and have adverse event data reported for both periods.
Arm/Group | Severe Renal Insufficiency Participants: Part 1 | Moderate Renal Insufficiency Participants: Part 1 | Healthy Control Participants: Part 1 | Severe Renal Insufficiency Participants: Part 2 | Moderate Renal Insufficiency Participants: Part 2 | Healthy Control Participants: Part 2
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/8 | 2/8 | 2/8 | 1/6 | 2/6 | 0/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Severe Renal Insufficiency Participants: Part 1 (N=8) | Moderate Renal Insufficiency Participants: Part 1 (N=8) | Healthy Control Participants: Part 1 (N=8) | Severe Renal Insufficiency Participants: Part 2 (N=6) | Moderate Renal Insufficiency Participants: Part 2 (N=6) | Healthy Control Participants: Part 2 (N=6)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site extravasation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypoaethesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.